CLINICAL TRIAL: NCT06622928
Title: Ventriculo-arterial Coupling in Patients With End-stage Renal Disease on Hemodyalisis: Intra-dialytic Changes and Prognostic Value.
Brief Title: Ventriculo-Arterial Coupling and Intra-Dialytic Changes in Hemodialysis Patients: Prognostic Insights
Status: Not yet recruiting | Type: Observational
Sponsor: Nazarbayev University (Other)
Collaborators: B.B.NURA, Center of efferent therapy and hemodialysis in Astana (Unknown); JSC National Research Cardiac Surgery Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: AP23490021
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis; Ventriculo-arterial Coupling
Keywords: hemodialysis; end-stage renal disease; ventriculo-arterial coupling; advanced echocardiography; cardiac ultrasound
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End-Stage Renal Disease Patients on Hemodialysis: Patients with end-stage renal disease (ESRD) undergoing regular hemodialysis, recruited based on specific inclusion and exclusion criteria. Inclusion criteria include patients aged 18 or older, receiving a standard renal replacement therapy of three dialysis sessions per week, with a dialysis history of at least 3 months and dialysis adequacy (Kt/V >1.2). Exclusion criteria include patients with a history of kidney transplantation, recent myocardial infarction or stroke, severe heart failure, chronic atrial fibrillation, obesity (BMI >40 kg/m²), and malignancy.
  Patients will undergo echocardiographic evaluations before and after dialysis, with a focus on left ventricular function and ventriculo-arterial coupling (VAC) using speckle-tracking echocardiography and pressure-volume loop analysis.
  Interventions: Diagnostic Test: Echocardiogram

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Echocardiographic Assessments:
  Pre-Hemodialysis Echocardiography:
  Before each hemodialysis session, echocardiograms will be performed to evaluate cardiac function and gather baseline data on ventriculo-arterial coupling (VAC) parameters. This will include recording three apical echocardiographic views (4-chamber, 2-chamber, and 3-chamber) by a trained sonographer.
  Post-Hemodialysis Echocardiography:
  Following the completion of the hemodialysis session, echocardiographic assessments will be repeated to measure changes in VAC parameters and other relevant cardiac metrics.

SUMMARY:
The acute effect of hemodialysis (HD) on left ventricular mechanics has been evaluated in several studies, however their results are not uniform. Eventually, the heart and the arterial system behave as an interconnected system and not as isolated structures; thus, the evaluation of the interaction of cardiac contractility with the arterial system would provide a more comprehensive understanding of the cardiovascular function and cardiac energetics. However, there have not been any studies demonstrating changes in terms of volumes, contractility, intraventricular pressure gradients distribution, and vascular properties in response to changes in loading conditions and their impact on the outcome.

With these concepts in mind, we aim to evaluate the effect of volume changes induced by HD on ventriculo-arterial coupling (VAC) computed from speckle-tracking echocardiography. In particular, we seek to study patients with end-stage renal disease (ESRD) to assess:

1. VAC parameters before and after the hemodialysis session;
2. The value of VAC parameters in predicting adverse outcome

Three-hundred-eighty-four patients with ESRD will be evaluated by standard 2-D echocardiography before and after the HD session. Echocardiographic speckle tracking images will be analysed off-line using a dedicated software based on a mathematical model (QStrain, Medis BV, Leiden, NL). The software reconstructs the pressure/volume (PV) loop by determining the end-systolic and end-diastolic pressure-volume relationship using the single-beat algorithms. The PV relation will be depicted for the entire cardiac cycle where each point of the curve is described as (Vt, Pt). Based on this integrated PV loop analysis, the following hemodynamic parameters will be calculated: LV systolic elastance (Ees); Arterial elastance (Ea); Ventricular-Arterial Coupling (VAC); Stroke Work (SW); Pressure-volume area (PVA); Work efficiency (WE).

Patients will be followed-up for 18 months. Primary end-point will be a composite of all-cause of death, nonfatal myocardial infarction, and hospitalization due to worsening heart failure. Secondary end-point will be a composite of cardiac death, nonfatal myocardial infarction, and hospitalization for heart failure. Event-free survival for each of the echocardiographic and VAC parameters will be assessed using Kaplan-Meier analysis and compared with a log-rank test, where each index will be dichotomized according to the median of its distribution. The prognostic value will be determined using the Cox proportional hazards model. Differences will be considered statistically significant when p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Standard renal replacement schedule with 3 dialysis sessions per week;
* Dialysis vintage of at least 3 months;
* Dialysis adequacy with single-pool Kt/V >1.2

Exclusion Criteria:

* Previous kidney transplantation
* Myocardial infarction, unstable angina or stroke during the previous 6 months;
* Severe stage III to IV congestive heart failure according to the NYHA classification;
* Chronic atrial fibrillation or other known arrhythmia;
* History of non-adherence to the prescribed weekly dialysis schedule in the previous month;
* Body mass index >40 Kg/m2; or
* History of malignancy or other clinical conditions associated with very poor prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 384 patients with end-stage renal disease (ESRD) recruited from the B.B. NURA Center of Efferent Therapy and Hemodialysis in Astana. This center, operational since 1988, provides comprehensive hemodialysis services, including 24/7 emergency care for patients requiring renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Interdialytic Changes in Ventricular-Arterial Coupling (VAC) and Its Prognostic Value in Patients Undergoing Regular Hemodialysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Salustri, MD, PhD, Principal Investigator — Nazarbayev University School of Medicine
Locations (1):
- Nazarbayev University School of Medicine, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bansal N, Zelnick L, Bhat Z, Dobre M, He J, Lash J, Jaar B, Mehta R, Raj D, Rincon-Choles H, Saunders M, Schrauben S, Weir M, Wright J, Go AS; CRIC Study Investigators. Burden and Outcomes of Heart Failure Hospitalizations in Adults With Chronic Kidney Disease. J Am Coll Cardiol. 2019 Jun 4;73(21):2691-2700. doi: 10.1016/j.jacc.2019.02.071. PMID 31146814
- [Background] Iseki K, Fukiyama K. Long-term prognosis and incidence of acute myocardial infarction in patients on chronic hemodialysis. The Okinawa Dialysis Study Group. Am J Kidney Dis. 2000 Oct;36(4):820-5. doi: 10.1053/ajkd.2000.17676. PMID 11007686
- [Background] Inuzuka R, Kass DA, Senzaki H. Novel, single-beat approach for determining both end-systolic pressure-dimension relationship and preload recruitable stroke work. Open Heart. 2016 Jun 15;3(1):e000451. doi: 10.1136/openhrt-2016-000451. eCollection 2016. PMID 27347424
- [Background] Zuo ML, Chen QY, Pu L, Shi L, Wu D, Li H, Luo X, Yin LX, Siu CW, Hong DQ, Gan H. Impact of Hemodialysis on Left Ventricular-Arterial Coupling in End-Stage Renal Disease Patients. Blood Purif. 2023;52(7-8):702-711. doi: 10.1159/000531188. Epub 2023 Aug 14. PMID 37579725
- [Background] Sasso L, Capuano A, Minco M, Paglia A, Pirozzi F, Memoli B, Carlomagno G, Petretta M, Bonaduce D. Hemodialysis does not affect ventricular-arterial coupling beyond the reduction of blood pressure and preload. Int J Cardiol. 2013 Sep 30;168(2):1553-4. doi: 10.1016/j.ijcard.2012.12.024. Epub 2013 Feb 27. No abstract available. PMID 23453441
- [Derived] Salustri A, Tonti G, Pedrizzetti G, Zhankorazova A, Khamitova Z, Toktarbay B, Jumadilova D, Khvan M, Galiyeva D, Bekbossynova M, Mukarov M, Kokoshko A, Gaipov A. Intradialytic Changes and Prognostic Value of Ventriculo-Arterial Coupling in Patients With End-Stage Renal Disease: Protocol for an Observational Prospective Trial. JMIR Res Protoc. 2025 Jun 23;14:e71948. doi: 10.2196/71948. PMID 40550123